CLINICAL TRIAL: NCT04400461
Title: Short-term Physical Function Outcomes in Severe COVID-19 Patients Admitted to ICU for Invasive Mechanical Ventilation: an Observational Cohort Study
Brief Title: Short-term Physical Function Outcomes in Severe COVID-19 Patients Admitted to ICU for Invasive Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Maria Natividad Seisdedos Nunez, Physiotherapist, MSc, Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Other Study IDs: 165/20
Record Dates: First submitted 2020-05-20; First posted 2020-05-22 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
Keywords: physical function; functional outcomes; strength; intensive care unit; rehabilitation
MeSH Terms: conditions — COVID-19 | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection and clinical testing of subjects — Clinical Testing: muscle strength. Muscle strength, as a component of physical function, will be assessed with the Medical Research Council sum score (MRC- SS) at discharge from the ICU and at discharge from the hospital.
  Clinical testing: physical function. The Functional Status Score for the ICU (FSS-ICU) will be used to evaluate 5 functional tasks at discharge from hospital.

SUMMARY:
Little is known about the physical function outcomes in patients with severe COVID-19 patients who are admitted to Intensive Care Unit (ICU) for invasive mechanical ventilation. The purpose of this study is to evaluate the short-term impact on physical function before hospital discharge in subjects with severe COVID-19 who have survived ICU admission for invasive mechanical ventilation.

DETAILED DESCRIPTION:
DESIGN: An observation cohort study conducted in a tertiary hospital.

METHODS: Data will be collected from patients along the ICU-hospital discharge continuum, will be analysed and non-parametric tests will be used to explore association between variables.

Outcome measures: Muscle strength, as a component of physical function, will be evaluated with the Medical Research Council sum score (MRC- SS) at discharge from ICU and at hospital discharge; the Functional Status Score for the ICU (FSS-ICU) will also be assessed at hospital discharge. Data on participants' demographics, ICU admission and hospital admission will also be collected.

SIGNIFICANCE OF THE RESEARCH: Understanding how physical function is affected in patients with severe COVID-19 may help develop future prevention, therapeutic and follow-up strategies that improve quality of care and outcomes in this specific group of patients. Findings from this study may be useful to design future larger cohort studies and experimental trials.

ELIGIBILITY:
Inclusion Criteria:

* subjects diagnosed with COVID-19 who have required admission to ICU for invasive mechanical ventilation;
* have received invasive ventilation > 24 hours;
* have been successfully weaned from mechanical ventilation > 48 hours;
* were independently able to mobilise prior to current hospital admission (this includes subjects who used a walking stick or another gait aid to mobilise.

Exclusion Criteria:

* subjects or proxies with inability to communicate in Spanish fluently;
* cognitive impairment prior to ICU admission;
* proven neurological impairment or neuromuscular disorder;
* Cerebrovascular Accident during hospital stay;
* previous organ transplant;
* pregnancy;
* unstable fractures or any other injuries that would require medical bed rest.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with COVID-19 who require admission to the ICU for invasive mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Medical Research Council sum score (MRC- SS). | < 48 hours before ICU discharge
  Physical examination will be performed to carry out manual muscle testing of strength in 6 different muscle groups of the upper limb and lower limb on both sides of the body.
Medical Research Council sum score (MRC- SS). | < 24 hours before hospital discharge
  Physical examination will be performed to carry out manual muscle testing of strength in 6 different muscle groups of the upper limb and lower limb on both sides of the body.
The Functional Status Score for the ICU (FSS-ICU) | < 24 hours before hospital discharge
  The Functional Status Score for the ICU (FSS-ICU) will be used to evaluate 5 functional tasks. Each task is evaluated using an 8-point ordinal scale ranging from 0 (not able to perform) to 7 (complete independence).The total FSS-ICU score ranges from 0 to 35, with higher scores indicating better physical functioning.

SECONDARY OUTCOMES:
Age | Through study completion, up to 6 months
  Age in years
Sex | Throughout study completion , up to 6 month
  Male vs Female
Body Mass Index | Throughout study completion, up to 6 months
  kg/m2
Baseline mobility | First day the patient can cooperate with assessment according to the ' 5 Standard Questions' test.
  Baseline mobility
APACHE II score | <24 hours after ICU admission
  Acute Physiology and Chronic Health Evaluation II score.The APACHE II score ranges from 0 to 71 points. Higher scores correspond to more severe disease and a higher risk of death.
Length of stay in ICU | Throughout the study completion, up to 6 months
  Number of days of stay in ICU
Number of days on mechanical ventilation | Throughout the study completion, up to 6 months
  Number of days on mechanical ventilation
Polyneuropathy diagnosis | Throughout the study completion, up to 6 months
  Clinical or EMG polyneuropathy diagnosis confirmation
Number of days on Neuromuscular Blockers | Throughout the study completion, up to 6 months
  Number of days on NMB during mechanical ventilation
Episodes of prone positioning | Throughout the study completion, up to 6 months
  Number of prone positioning episodes during ICU stay
Length of stay in hospital | Throughout the study completion, up to 6 months
  Total number of days admitted to hospital
Continuation of care | Throughout the study completion, up to 6 months
  Home with no follow-up physiotherapy, home with domiciliary or out-patient physiotherapy, rehabilitation facility, care home, transfer to another acute hospital.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Medical ICU. Hospital Universitario Ramón y Cajal, Madrid
  - Surgical ICU. Hospital Universitario Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No